CLINICAL TRIAL: NCT06460610
Title: Comparative Effects of Blow Bottle and Acapella Along With Diaphragmatic Breathing in Patients With Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0383
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Pneumonia
Keywords: blow bottle; acapella; diaphragmatic breathing; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blow Bottle technique (Experimental): Blow Bottle Technique will be performed to emphasizing deep diaphragmatic breathing and controlled exhalation. Blow Bottle sessions for up to 20 minutes per day for 3 days in a week .Total 12 sessions in 4 weeks.
  Interventions: Other: Blow Bottle technique
- (Acapella along with Diaphragmatic Breathing) (Active Comparator): Acapella will be performed to Improves clearance of secretion to facilitates opening of airway in patients with lung disease to mobilize secretions and improve lung function. Daily session for 20 minutes per day for 3 days in a week. Total 12 sessions in 4 weeks
  Interventions: Other: Acapella along with Diaphragmatic Breathing

INTERVENTIONS:
Other: Blow Bottle technique — Patients sit at a table with comfortable position Hold the bottle with one hand and the tube with the other Put the tube in mouth by holding lips firmly Breath in through nose and out through mouth Blowing enough water is bubbled Short Breaks for 2 to 3 mints When mucus rises up get out of it by coughing or huffing
  Arms: Blow Bottle technique
Other: Acapella along with Diaphragmatic Breathing — Device which uses a counter weighted plug and magnet to create airway oscillations Acapella combines the effects of PEP therapy and airway vibrations and mobilize to clear pulmonary secretions Facilitates opening of airways in patients with lung disease. Patients instructions to close the mouth piece making surety to no leakage of air. Take a long breath in nose and blow out through the Acapella ,feel vibrations on chest. Duration of performing this technique 3 days a week for 20 mints per day, 4 weeks regular
  Arms: (Acapella along with Diaphragmatic Breathing)

SUMMARY:
Pneumonia is the inflammation of lung parenchyma involving lungs alveoli and is a leading cause of lower respiratory tract infections and deaths around the globe and the number rises greatly after the Covid-19 pandemic. The Symptoms of Pneumonia is cough, fever, dyspnea, myalgia, altered blood gas ratio, and mental alteration. Treatment and management of this disease varies from patient to patient according to its severity stages .Blow Bottle supports the patient to remove excess secretions to increase pressure in the airways. This opens up the passageways in bronchioles, air behind the mucus push it into the larger airways .It will be easy to remove mucus by coughing or huffing. Hypoximia is a clinical feature of Pneumonia that requires a fraction of inspired oxygen FiO2 of 0.50 to maintain an oxygen saturation of 92%. This research of randomized clinical trial will check the comparative effects of Blow Bottle Technique and Acapella along with Diaphragmatic Breathing in patients with Pneumonia by taking sample of 50 patients through Non Probability convenience sampling and randomly allocating them to two groups A and B out of which A will receive both Blow Bottle and Diaphragmatic Breathing training, B will receive Acapella with Diaphragmatic Breathing upto the duration of 3 days per week for upto 4 weeks. Pre and post training outcomes of pulmonary function will be measured through BCSS ,Oxygen Saturation through Pulse Oximeter, and disease severity through Pneumonia severity index, and Who QOL questionnaire. The data will be analyzed through SPSS 21

ELIGIBILITY:
Inclusion Criteria:

* Patients in the acute pneumonia
* Age40-60 years.
* Both male and female
* Patients with unstable health conditions
* Participants were willing to participate

Exclusion Criteria:

* Patients with physical or cognitive limitations.
* Patients with a history of chronic respiratory conditions such as COPD, bronchitis, or asthma
* Pregnant or breastfeeding women. Individuals with musculoskeletal or neurological conditions
* Patients with contraindications to chest percussion therapy, such as recent surgery or trauma to the chest area.
* Patients with severe Pneumonia requiring immediate care

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Pulse Oximeter | baseline and fourth week
  Pulse oximetry is a noninvasive test that measures the oxygen saturation level of your blood
Who QOL Questionnaire | baseline and fourth week
  Quality of life Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale The physical health domain includes items on mobility, daily activities, functional capacity, energy, pain, and sleep.
Breathlessness, Cough and Sputum Scale | baseline and fourth week
  The Breathlessness, Cough and Sputum Scale (BCSS) is used to predict patient exacerbations by evaluating common symptoms identified in the COPD population. The BCSS have 24 items concerning beliefs about the self and others that are assessed on a five-point rating scale (0-4).Four scores are obtained: negative-self (six items), positiveself (six items), negative-others (six items) and positive-others (six items)

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres A, Chalmers JD, Dela Cruz CS, Dominedo C, Kollef M, Martin-Loeches I, Niederman M, Wunderink RG. Challenges in severe community-acquired pneumonia: a point-of-view review. Intensive Care Med. 2019 Feb;45(2):159-171. doi: 10.1007/s00134-019-05519-y. Epub 2019 Jan 31. PMID 30706119
- [Background] Quinton LJ, Walkey AJ, Mizgerd JP. Integrative Physiology of Pneumonia. Physiol Rev. 2018 Jul 1;98(3):1417-1464. doi: 10.1152/physrev.00032.2017. PMID 29767563